CLINICAL TRIAL: NCT00069589
Title: Alopecia Areata Registry and Immunogenetic Mechanisms
Brief Title: Alopecia Areata Registry
Acronym: NAAR
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Alopecia Areata Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NIAMS-097; HHSN268200682279C; NCT00177073 (obsolete NCT alias)
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis; Autoimmune Hair Loss; Alopecia Partialis
Keywords: Baldness; Autoimmunity; Hair; Alopecia Areata; Alopecia Partialis; Alopecia Totalis; Alopecia Universalis; Autoimmune Hair Loss
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Alopecia; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be analyzed to learn the link between gene markers of traites of alopecia areata. Sera will be used to analyse cytokins. Lymphocytes will be used for the creation of B-cell lines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alopecia areata is the loss of hair in patches that can proceed to loss of all hair (alopecia totalis or universalis). The purpose of the registry is to collect patient information and blood samples from people with alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata is a condition in which hair is lost either from part of the scalp, all of the scalp, or the entire body, and it affects 1% to 2% of the population. It is thought to be an autoimmune disease and in some cases the disease is hereditary. The Alopecia Areata Registry will collect information and blood samples from clinically well-characterized patients with these three forms of alopecia areata: alopecia partialis (patchy loss of the scalp hair), alopecia totalis (total loss of all scalp hair), and alopecia universalis (complete loss of all hair everywhere on the body). This will be a collection of patients in multi-generational families, twins, single patients with patchy, persistent transient alopecia areata or long-standing alopecia totalis/universalis and with controls (persons unaffected and not related to alopecia patients). Information from these patients will be used to search the human genome for disease-associated loci and/or genes. Researchers interested in doing pathophysiology or treatment studies of this disease will also be able to contact patients having the appropriate form of the disease for the studies in question.

Patients who have been diagnosed with alopecia areata by a dermatologist will be eligible for the registry. Patients will fill out an information form online (alopeciaareataregistry.org). Patients who have a family history or specific types of alopecia will be invited to participate in a more detailed questionnaire and physical exam and have blood samples drawn.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with alopecia areata by a dermatologist
* United States resident

Accepts Health Volunteers: Non blood-related individuals who are unaffected with alopecia areata and do not live in the same household with alopecia areata patient.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with alopecia areata (AA), both children and adults, who have been diagnosed by a physician with alopecia universalis, alopecia totalis, patchy persistent AA, or transient mild AA. Family members (related by blood) of these patients, preferably sib-pairs plus parents and multiplex families(persons with at least three family members with AA or alopecia universalis and alopecia totalis).
  Also, healthy individuals who are unaffected, non-blood related individuals and do not live in the same household with alopecia areata patient are needed as controls.
Sampling Method: Probability Sample
Enrollment: 3100 (Estimated)
Dates: Start 2001-11; Primary Completion 2099-11 (Estimated); Study Completion 2099-11 (Estimated)

PRIMARY OUTCOMES:
Alopecia Areata Registry | Registration on-going
  Database registration of participants via collection of participant epidemiology data.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Duvic, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado - UCHSC - Health Science Center at Fitzsimons, Aurora, Colorado
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Duvic M, Norris D, Christiano A, Hordinsky M, Price V. Alopecia areata registry: an overview. J Investig Dermatol Symp Proc. 2003 Oct;8(2):219-21. doi: 10.1046/j.1087-0024.2003.00814.x. PMID 14582678
- [Result] Barahmani N, Yang Y, Lopez A, Duvic M. Atopic alopecia areata patients have increased serum Th1 Cytokine profiles. 66th Annual meeting of Society for Investigative Dermatology. St.Louis, MO, May 2005. JID 124 (4): A100, 2005.
- [Result] Breuer-McHam J, Hunzicker K, Barahmani N, Zhang Q, Babu D, Christiano A, Hordinsky M, Norris D, Price V, Duvic, M. Epidemiologic and disease associations in participants of the national alopecia areata (NAAR) registrants. Accepted by Society for Investigational Dermatology, April 12, 2004. JID 122 (3): A107, 2004.
- [Result] de Andrade M, Barahmani N, Hunzicker K, Zhang Q, Joan Breuer- McHam, Joyce Osei, Daniel Babu, Qingyi Wei, Reveille J, Duvic M. HLA Class II associations confirm alopecia areata phenotypic subsets. 66th Annual meeting of Society for Investigative Dermatology. St. Louis, MO, May 2005.JID 124 (4): A107, 2005.
- [Result] Barahmani N, de Andrade M, Slusser JP, Wei Q, Hordinsky M, Price VH, Christiano A, Norris D, Reveille J, Duvic M. Human leukocyte antigen class II alleles are associated with risk of alopecia areata. J Invest Dermatol. 2008 Jan;128(1):240-3. doi: 10.1038/sj.jid.5700973. Epub 2007 Jul 19. No abstract available. PMID 17637820
- [Result] Ahmed AM, Barahmani N, Duvic M; National Alopecia Areata Registry. Familial alopecia areata and chronic thrombocytopenia. J Am Acad Dermatol. 2008 May;58(5 Suppl 1):S75-7. doi: 10.1016/j.jaad.2007.05.017. PMID 18489053
- [Result] Rodriguez TA, Duvic M; National Alopecia Areata Registry. Onset of alopecia areata after Epstein-Barr virus infectious mononucleosis. J Am Acad Dermatol. 2008 Jul;59(1):137-9. doi: 10.1016/j.jaad.2008.02.005. Epub 2008 Mar 7. PMID 18329131
- [Result] Martinez-Mir A, Zlotogorski A, Gordon D, Petukhova L, Mo J, Gilliam TC, Londono D, Haynes C, Ott J, Hordinsky M, Nanova K, Norris D, Price V, Duvic M, Christiano AM. Genomewide scan for linkage reveals evidence of several susceptibility loci for alopecia areata. Am J Hum Genet. 2007 Feb;80(2):316-28. doi: 10.1086/511442. Epub 2007 Jan 5. PMID 17236136
- [Result] Barahmani N, de Andrade M, Slusser JP, Zhang Q, Duvic M. Major histocompatibility complex class I chain-related gene A polymorphisms and extended haplotypes are associated with familial alopecia areata. J Invest Dermatol. 2006 Jan;126(1):74-8. doi: 10.1038/sj.jid.5700009. PMID 16417220
- See also: National Alopecia Areata Foundation (NAAF) official website — http://www.naaf.org